CLINICAL TRIAL: NCT01231113
Title: Efficacy, Safety and Tolerability of Dihydroartemisinin-Piperaquine for Treatment of Uncomplicated Falciparum Malaria in Pregnancy: an Open-label, Randomised Controlled, Non-inferiority Trial
Brief Title: Efficacy,Safety and Tolerability of Dihydroartemisinin-Piperaquine for Uncomplicated Malaria in Pregnancy in Ghana
Acronym: DHAPPQ/MIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kwame Nkrumah University of Science and Technology (Other)
Collaborators: Malaria Capacity Development Consortium (Unknown)
Responsible Party: Principal Investigator, Joseph Osarfo, Principal Investigator, Kwame Nkrumah University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 8/DHAPPQ/MIP
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Pregnancy Complicated by Malaria as Antepartum Condition
Keywords: malaria,; pregnancy,; dihydroartemisinin-piperaquine,; efficacy,; safety,; Ghana
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- artesunate-amodiaquine arm (Active Comparator): A co-blistered pack of amodiaquine and artesunate.The 452 pregnant women in this arm will receive artesunate-amodiaquine tablets(artesunate 4mg/kg and amodiaquine 10mg/kg in twelve hourly doses over 3 days
  Interventions: Drug: artesunate-amodiaquine
- Dihydroartemisinin-piperaquine arm (Experimental): a fixed-dose combination to be administered to the other 452 pregnant women in this arm at an estimated total dosing of 6.75mg/kg dihydroartemisinin and 55mg/kg piperaquine over 3 days
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: artesunate-amodiaquine — The 452 pregnant women in this arm will receive artesunate-amodiaquine tablets(artesunate 4mg/kg and amodiaquine 10mg/kg in twelve hourly doses over 3 days
  Other Names: camosunate
  Arms: artesunate-amodiaquine arm
Drug: Dihydroartemisinin-piperaquine — a fixed-dose combination to be administered to the other 452 pregnant women in this arm at an estimated total dosing of 6.75mg/kg dihydroartemisinin and 55mg/kg piperaquine over 3 days
  Other Names: artekin
  Arms: Dihydroartemisinin-piperaquine arm

SUMMARY:
Malaria in pregnancy poses enormous public health challenges, contributing to significant maternal and infant deaths yearly. Adverse outcomes include maternal anaemia and low birthweight. Down regulation of cellular immunity increases pregnant women's susceptibility to malaria and mediate these adverse outcomes.

The World Health Organization recommends treatment with artemisinin-combination therapy. Ghana uses quinine for malaria in first trimester pregnancies while artesunate-amodiaquine (AS-AQ) and quinine again are used in later trimesters. Recent amendments added artesunate-lumefantrine and dihydroartemisinin-piperaquine (DHA-PPQ) to the antimalarials used in the country. A high degree of safety and efficacy of DHA-PPQ is documented in several studies. DHA-PPQ, though not specified for use in pregnancy as of now, is accessible and available following its inclusion in the national malaria guidelines and may inadvertently be used to treat malaria in pregnancy. Paucity of data on DHA-PPQ use in pregnancy makes it pertinent to study its safety, tolerability and efficacy in pregnancy.

We propose an open label, randomized controlled non-inferiority comparison of DHA-PPQ and AS-AQ for treatment of uncomplicated malaria in pregnancy in second and third trimesters to assess safety, tolerability and efficacy of DHA-PPQ. Outcomes of interest include PCR-corrected cure rates at days 28 and 42, maternal haemoglobin levels at days 14 and 42, prevalence of congenital abnormalities and pregnancy wastage. Proportions and percentages will be described at 95% Confidence Intervals and compared using chi-square tests. Parametric and non-parametric tests of significance will be applied as appropriate to determine significance of differences in outcomes between the treatment groups.

DETAILED DESCRIPTION:
Pregnant women of all ages, gravidity and with gestational ages 16-30 weeks, living within 15 km of the study center and presenting for antenatal care or diagnosed with uncomplicated malaria will be screened with P.falciparum rapid diagnostic test kits after obtaining consent. Those testing positive will have blood film microscopy done and only those with positive blood film microscopy will be recruited to participate in the study. Participants will be randomized to receive either dihydroartemisinin-piperaquine at an estimated total dosing of 6.75mg/kg of dihydroartemisinin and 55mg/kg of piperaquine for 3 days rounded to the nearest half tablet) or artesunate-amodiaquine(artesunate 4mg/kg and amodiaquine 10mg/kg in two twelve hourly doses daily for 3 days) after giving informed consent and a physical examination. This will be followed by home visits on days 1, 3, 7, 14, 28 and 42 post-treatment to assess occurrence of adverse events and to obtain blood samples for microscopy, filter paper blots for PCR analysis and haematology. The mentioned laboratory investigations will also be conducted at recruitment.

Participants will be followed up to delivery and 6 weeks post-partum to gather data on maternal peripheral and placental parasitaemia, cord parasitaemia, maternal haemoglobin levels, low birth weights, stillbirths, preterm deliveries, neonatal jaundice, birth defects and infant deaths.

ELIGIBILITY:
Inclusion Criteria:

* RDT positive + microscopy confirmed P. falciparum parasitaemia. ii) Informed consent. iii) Resident within the defined 15km radius of the study center. iv) No history of antimalarial treatment in the preceding two weeks. v) Assurance of adherence to study requirements, follow-up and delivery at the hospital.

vi) Haemoglobin ≥ 7g/dl.

Exclusion Criteria:

* i) Confirmed multiple gestation. ii) Severe malaria or disease likely to influence pregnancy outcome eg renal/ cardiac disease, diabetes mellitus, known pregnancy induced hypertension, known human immunodeficiency virus infection.

iii) Known allergies to study medication. iv) Antimalarial treatment administered by a third party during the follow-up.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 417 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
PCR-corrected parasitological cure rates at days 28 and 42 | 42-day follow-up
  Only eligible subjects with positive falciparum rapid diagnostic test results and positive blood films on microscopy will be recruited. Filter paper blots will be prepared at recruitment as well.
  Blood films and filter paper blots will be repeated on days 3,7,14,28 and 42 post-first dose of treatment.
  PCR analysis will be conducted on only those follow-ups with positive blood films

SECONDARY OUTCOMES:
prevalence of birth defects | assessment made 24-72 hours post-partum
  birth defects obvious on inspection
Comparative prevalence of adverse and serious adverse events | three-monthly and at end of study
  the data monitoring committee will assess adverse events data quarterly and advice accordingly. Where there is no justification to stop the study before completion, the final assessments will done on study completion
pregnancy outcomes (spontaneous abortions, still births, preterm delivery, etc) | quaterly from first recorded delivery and on completion
  data monitoring committee will assess generated data on the above and advice accordingly

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Osarfo, MBCHB, MPH, Principal Investigator — Malaria Capacity Development Consortium-Ghana, Department of Community Health, School of Medical Science, Kwame Nkrumah University of Science and Technology; Harry Tagbor, PhD, Study Director — Kwame Nkrumah University of Science and Technology; Pascal Magnussen, Study Director — DBL-University of Copenhagen
Locations (1):
- St.Michael's Hospital, Pramso, Kumasi, Ashanti Region, Ghana